CLINICAL TRIAL: NCT00491803
Title: Acute Effects of a Single Dose of Sildenafil (20mg/40mg) on Pulmonary Haemodynamics and Gas Exchange at Rest and During Exercise in COPD Patients With Pulmonary Hypertension
Brief Title: Sildenafil Effects on Pulmonary Haemodynamics and Gas Exchange in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: SIL-COPD-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Joan Albert Barbera, Hospital Clinic Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIL-COPD-01; EudraCT #: 2007-000116-81
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sildenafil 20mg
  Interventions: Drug: Sildenafil
- 2 (Active Comparator): Sildenafil 40mg
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — sildenafil 20 mg orally
  Arms: 1
Drug: Sildenafil — sildenafil 40 mg orally
  Arms: 2

SUMMARY:
Sildenafil is a phosphodiesterase-5 inhibitor that has been approved for the treatment of pulmonary arterial hypertension with orphan drug designation. Sildenafil modulates the nitric oxide (NO) pathway in the vessel wall. Since this pathway is impaired in pulmonary arteries of patients with pulmonary hypertension (PH) associated with chronic obstructive pulmonary disease (COPD), we hypothesized that sildenafil might improve pulmonary hemodynamics and increase exercise tolerance in this condition. However, in COPD sildenafil may also impair gas exchange due to the inhibition of pulmonary hypoxic vasoconstriction. The research project is aimed to evaluate these effects.

It is a prospective, randomized, double-blind study to evaluate the acute effects of a single dose of 20 or 40 mg of sildenafil on gas exchange and pulmonary hemodynamics. Subjects: 20 patients (10 in each group). Measurements: pulmonary hemodynamics, arterial blood gasses and ventilation-perfusion distributions; at rest and during sub-maximal exercise.

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1/FVC<0.7)
* Age 40-75
* Pulmonary hypertension (Vmax TI>=2.8m/sec)

Exclusion Criteria:

* Treatment with CYP3A4 inhibitors, nitrates, PDE-5 inhibitors
* Coronary disease
* Ischemic optical neuritis

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Reduction of mean PAP and PVR | 60 minutes

SECONDARY OUTCOMES:
CO, PaO2, V/Q | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joan albert Barbera, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Blanco I, Gimeno E, Munoz PA, Pizarro S, Gistau C, Rodriguez-Roisin R, Roca J, Barbera JA. Hemodynamic and gas exchange effects of sildenafil in patients with chronic obstructive pulmonary disease and pulmonary hypertension. Am J Respir Crit Care Med. 2010 Feb 1;181(3):270-8. doi: 10.1164/rccm.200907-0988OC. Epub 2009 Oct 29. PMID 19875684